CLINICAL TRIAL: NCT03786497
Title: Protecting Brains and Saving Futures - the PBSF Protocol: a Prospective Multicenter and Observational Study on the Use of Telemedicine for Neurocritical Care in High-risk Newborns in Brazil.
Brief Title: Protecting Brains and Saving Futures - the PBSF Protocol
Acronym: PBSF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Protecting Brains Saving Futures (Other)
Responsible Party: Principal Investigator, Dr Gabriel Variane, Physician, Protecting Brains Saving Futures
Other Study IDs: PBSF_2020
Record Dates: First submitted 2018-12-12; First posted 2018-12-26 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Brain Injuries; Congenital Heart Disease; Newborn Morbidity; Intraventricular Hemorrhage; CNS Infection; Neonatal Seizure; Nosocomial Infection; Hypoxic-Ischemic Encephalopathy; Extreme Prematurity; Brain Malformation; Congenital Infection; Neonatal Stroke; Hemodynamic Instability; Extracorporeal Membrane Oxygenation Complication; Inborn Errors of Metabolism; Respiratory Complication; Neonatal Death
Keywords: Newborn; Neonatal Neurocritical Care Units; Neonatal Brain Monitoring; Brain Injury; Neuroprotection; Telemedicine; Electroencephalography; Amplitude-Integrated Electroencephalography; Near Infrared Spectroscopy; Neurodevelopmental Problems
MeSH Terms: conditions — Brain Injuries; Heart Defects, Congenital; Central Nervous System Infections; Cross Infection; Hypoxia-Ischemia, Brain; Metabolism, Inborn Errors; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Multiple neonatal disorders are associated with risks of neurological injury. Thus, management of these infants should involve a coordinated approach to permit early diagnosis with improved clinical care. Such initiative involves the use of standardized protocols, continuous and specialized brain monitoring with electroencephalography (EEG), amplitude integrated EEG (aEEG) and Near Infrared Spectroscopy (NIRS), neuroimaging and training. Brazil is a very large country with disparities in health care assessment; some neonatal intensive care units (NICUs) are not well structured and trained to provide adequate neurocritical care. However, the development and implementation of these neurocritical care units requires high expertise and significant investment of time, manpower and equipment. In order to reduce the existing gap, a unique advanced telemedicine model of neurocritical care called Protecting Brains and Saving Futures (PBSF) protocol was developed and implemented in some Brazilian NICUs.

Methods: A prospective observational cohort study will be conducted in 20 Brazilian NICUs that have adopted the PBSF protocol. All infants receiving the protocol during January 2021 to December 2023 will be eligible. Ethical approval will be obtained from the participating institutions. The primary objective is to describe the use of the PBSF protocol and clinical outcomes, by center and over a 3 years period. The use of the PBSF protocol will be measured by quantification of neuromonitoring, neuroimaging exams and sub-specialties consultation. Clinical outcomes of interest after the protocol implementation are length of hospital stay, detection of EEG seizures during hospitalization, use of anticonvulsants, inotropes, and fluid resuscitation, death before hospital discharge, and referral of patients to high-risk infant follow-up. These data will be also compared between infants with primarily neurologic and primarily clinical diagnosis.

Discussion: The implementation of the PBSF protocol may provide adequate remote neurocritical care in high-risk infants with optimization of clinical management and improved outcomes. Data from this large, prospective, multicenter study are essential to determine whether neonatal neurocritical units can improve outcomes. Finally, it may offer the necessary framework for larger scale implementation and help in the development of studies of remote neuromonitoring.

DETAILED DESCRIPTION:
METHODS Objectives The aim of this multicenter, prospective, cohort study is to describe the use of the PBSF protocol and clinical outcomes, by center and over a 3 years period (2021 to 2023) in the NICUs that have adopted it. We hypothesize that the use of the PBSF protocol will increase over time with improvement of some specific short-term outcomes (see methods below). Results of this study may provide the necessary background information for larger studies and initiatives aiming to protect neonatal brains and save futures.

Study Design and Setting This will be a multicenter, prospective, observational study in a cohort of high-risk neonates treated at 20 different NICU's in Brazil. The intended period of patient recruitment and data collection will be 3 years (January 2021 to December 2023). The study followed the precepts of good clinical practice and was approved by the Research Ethics Committee of the Irmandade da Santa Casa de Misericórdia de São Paulo. In addition, the project has received formal authorization from the Clinical and Administrative Board of each center. When selecting a participant, the principal investigator of the study or one of the co-investigators will contact the parents or guardians and obtain informed consent. All data will be treated anonymously and confidentially, and in no phase of the study any name, image, or data that allows participants identification will be disclosed.

Participants In this cohort study, all the infants admitted to any of the 20 NICUs from birth up to three months of life and receiving the PBSF protocol are eligible. Indications for the use of the protocol are provided on Box 1. Patients with genetic syndromes or malformation incompatible with life, or older than three months old will be excluded. Details on the PBSF protocol are provided in supplemental material. Briefly, the protocol includes provision of equipment and resources, connection between the associated NICU and the remote monitoring center called the Central of Surveillance and Intelligence (CSI), training and teaching of all health care professional team of each NICU, and customized multiparametric recordings of biological signals of each patient monitoring. At the CSI, a team is available 24 hours a day all year around, allowing for case discussions and simplified reports of brain monitoring information on the patient monitor's display every 6 hours.

Variables Population demographics: gender, gestational age at birth, gestational age ≤ 32 weeks and < 37 weeks, Apgar score at 1 min, 5 min and 10 min, birth weight, current weight, inborn or outborn, use of antenatal steroids and magnesium sulfate, type of birth.

Primary diagnosis: seizure, anoxia/mild HIE, moderate or severe HIE/cooling, neurologic abnormalities without specific diagnosis, congenital central nervous system (CNS) anomalies, grade III or IV intraventricular hemorrhage (IVH) or hydrocephalus, periventricular leukomalacia, meningitis, neural tube defects, stroke, cyanotic congenital heart defect (CHD), prematurity, gestational age ≤ 32 weeks, meconium aspiration syndrome, cardiorespiratory instability, necrotizing enterocolitis, metabolic disease, extracorporeal membrane oxygenation (ECMO)/pre-ECMO and any other medical conditions not listed here.

For descriptive analysis of the 2 main outcomes (use of the PBSF protocol and clinical outcomes) patients will be them divided into two groups accordingly to their primary diagnosis: neurological or clinical.

Data sources / measurement Patient demographics, diagnosis and clinical outcomes will be extracted from the medical charts of each patient enrolled and entered in the PBSF database. The use of the PBSF protocol will be measured with the data collected by the CSI center continuously. Details of these recordings are provided on Appendix 2.

Bias To address potential source of bias related to financial availability, the 2 main outcomes of interest will be also adjusted based on the unit primary profile: private, foundation or public.

Study size Based on our current experience, there are an average of 5 patients per month with criteria for neurocritical care on each center, making a total of 3,240 eligible patients during a three years period. Considering a 30% loss due to refusal to consent, non-availability of the research team or missing data, we expect to recruit 2,268 infants from all study centers (around 756 patients per year).

Statistical methods Categorical variables will be analyzed by descriptive statistics and presented as number of valid cases and percentage (%). Numeric variables will be analyzed as mean and standard deviation, median and interquartile ranges, or coefficient intervals. Chi-square test (or Fisher's exact test) will be performed to analyze categorical variables and the Student's t test, or Wilcoxon rank sum test will be used to check for significant differences between the two groups. A p value of <0.05 will be considered statistically significant. The confidence interval considered will be 95%. Analysis of variability (distribution) per site for each variable of the 2 main outcomes will also be performed. ANOVA with post hoc Bonferroni will be used to compare outcomes over time, i.e. between years 1, 2 and 3 and Kaplan Meier curves will be generated to follow the evolution of outcomes over time for the 2 groups of patients: neurologic and clinical.

Results Participants. A flow chart of all eligible and enrolled patients will be produced, and the total number of patients will be reported, overall and per center.

Descriptive data Population demographics: male, n (%); gestational age at birth, weeks, mean (SD); gestational age ≤ 32 wk, n(%); Gestational age < 37 wk, n (%); Apgar score at 1 min, at 5 min, and at 10min, median (IQR); birth weight, grams, mean (SD); current weight, grams, mean (SD); Inborn, n (%); use of antenatal steroids and magnesium sulfate, n (%); Caesarean, n(%).

Primary outcomes:

Use of the PBSF protocol

1. Use of aEEG/EEG monitoring
2. Duration of aEEG/EEG monitoring
3. Number primary neurologic or medical patients with aEEG or EEG monitoring and the duration of the monitoring (hours)
4. Number of primary neurologic or medical patients with NIRS monitoring and the duration of the NIRS monitoring (hours)
5. Number of primary neurologic or medical patients with brain MRI, neurology consult, and neurosurgery consult.
6. Number of clinical case discussions and videoconference meetings

Clinical outcomes

1. Length of hospital stay
2. Number of electroencephalographic seizures during hospitalization
3. Use and types of anticonvulsants administered
4. Number and types of anticonvulsants prescribed at discharge
5. Use and types of inotropes administered during NICU stay
6. Use and types of fluid resuscitation administered during NICU stay
7. Death before hospital discharge
8. Number of patients referred to neurology or neurosurgery
9. Number of patients referred to high-risk infant follow-up*

Secondary outcomes:

Use of the PBSF protocol

1. Number of remote communications between CSI and local team
2. Number of reports issued for aEEG / EEG exams with or without the use of NIRS
3. Number of patients who performed Therapeutic Hypothermia
4. Association of pathological brain monitoring findings (aEEG/EEG and NIRS) and alterations in imaging exams including brain magnetic resonance imaging (brain MRI) and cranial ultrasonography (cranial US) performed during hospitalization
5. Association of pathological brain monitoring findings with morbi-mortality and length of hospital stay
6. Adverse effects of therapeutic hypothermia measured by cardiac arrhythmia, thrombocytopenia and coagulation disorders in general, skin lesion and pulmonary hypertension
7. Adverse effects of brain monitoring expressed by skin lesion due to electrode / sensor positioning
8. Association of pathological brain monitoring findings with evaluation of neurodevelopment by application of the Bayley test between 18 and 24 months of life

ELIGIBILITY:
- Inclusion criteria:

In this cohort study, all the infants admitted to any of the 20 NICUs from birth up to three months of life and receiving the PBSF protocol are eligible. Following are the indications for use of the PBSF protocol in the participating centers

1. Extreme prematurity
2. Peri-intraventricular Hemorrhage
3. Hypoxic-ischemic encephalopathy (mild, moderate or severe)
4. Congenital heart disease
5. Neonatal stroke
6. Congenital infections
7. Nosocomial infections
8. Inborn errors of metabolism
9. Severe hemodynamic/ventilatory instability
10. Seizures
11. Brain malformations
12. CNS infection
13. ECMO

    * Exclusion criteria:

Patients with genetic syndromes or malformation incompatible with life, or older than three months old will be excluded.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This will be a multicenter, prospective, observational study in a cohort of high-risk neonates treated at 20 different Neonatal Intensive Care Units in terciary hospitals in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 2268 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Applicability of telemedicine model for monitored infants | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Applicability of telemedicine model for recorded remote monitoring | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Use of aEEG/EEG monitoring | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Duration of aEEG/EEG monitoring | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number primary neurologic or medical patients with aEEG or EEG monitoring and the duration of the monitoring (hours) | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of primary neurologic or medical patients with NIRS monitoring and the duration of the NIRS monitoring (hours) | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of primary neurologic or medical patients with brain MRI, neurology consult, and neurosurgery consult. | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of clinical case discussions and videoconference meetings | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Length of hospital stay | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of electroencephalographic seizures during hospitalization | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Use and types of anticonvulsants administered | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number and types of anticonvulsants prescribed at discharge | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Use and types of inotropes administered during NICU stay | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Use and types of fluid resuscitation administered during NICU stay | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Death before hospital discharge | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of patients referred to neurology or neurosurgery | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of patients referred to high-risk infant follow-up | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).

SECONDARY OUTCOMES:
Number of remote communications between CSI and local team | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of reports issued for aEEG / EEG exams with or without the use of NIRS | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Number of patients who performed Therapeutic Hypothermia | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Association of pathological brain monitoring findings (aEEG/EEG and NIRS) and alterations in imaging exams including brain magnetic resonance imaging (brain MRI) and cranial ultrasonography (cranial US) performed during hospitalization | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Association of pathological brain monitoring findings with morbi-mortality and length of hospital stay | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Adverse effects of therapeutic hypothermia measured by cardiac arrhythmia, thrombocytopenia and coagulation disorders in general, skin lesion and pulmonary hypertension | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Adverse effects of brain monitoring expressed by skin lesion due to electrode / sensor positioning | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).
Association of pathological brain monitoring findings with evaluation of neurodevelopment by application of the Bayley test between 18 and 24 months of life | 3 years period
  Each outcome for all sites together will be also compared for changes over time from Year 1 (2021) to Year 3 (2023).

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Sant'Anna, PhD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Brazil (2):
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo
  - Protecting Brains and Saving Futures - PBSF, São Paulo

REFERENCES:
- [Background] Kurinczuk JJ, White-Koning M, Badawi N. Epidemiology of neonatal encephalopathy and hypoxic-ischaemic encephalopathy. Early Hum Dev. 2010 Jun;86(6):329-38. doi: 10.1016/j.earlhumdev.2010.05.010. Epub 2010 Jun 16. PMID 20554402
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Lawn JE, Wilczynska-Ketende K, Cousens SN. Estimating the causes of 4 million neonatal deaths in the year 2000. Int J Epidemiol. 2006 Jun;35(3):706-18. doi: 10.1093/ije/dyl043. Epub 2006 Mar 23. PMID 16556647
- [Background] Shankaran S, Woldt E, Koepke T, Bedard MP, Nandyal R. Acute neonatal morbidity and long-term central nervous system sequelae of perinatal asphyxia in term infants. Early Hum Dev. 1991 May;25(2):135-48. doi: 10.1016/0378-3782(91)90191-5. PMID 1713544
- [Background] Robertson CMT. Long-term follow-up of term infants with perinatal asphyxia. In: Stevenson DK, Benitz WE, Sunshine P. Fetal and neonatal brain injury. 3. Ed. New York: Cambridge University; 2003. p.829-58.
- [Background] de Vries LS, Jongmans MJ. Long-term outcome after neonatal hypoxic-ischaemic encephalopathy. Arch Dis Child Fetal Neonatal Ed. 2010 May;95(3):F220-4. doi: 10.1136/adc.2008.148205. PMID 20444814
- [Background] Marlow N, Rose AS, Rands CE, Draper ES. Neuropsychological and educational problems at school age associated with neonatal encephalopathy. Arch Dis Child Fetal Neonatal Ed. 2005 Sep;90(5):F380-7. doi: 10.1136/adc.2004.067520. PMID 16113154
- [Background] Blencowe H, Lee AC, Cousens S, Bahalim A, Narwal R, Zhong N, Chou D, Say L, Modi N, Katz J, Vos T, Marlow N, Lawn JE. Preterm birth-associated neurodevelopmental impairment estimates at regional and global levels for 2010. Pediatr Res. 2013 Dec;74 Suppl 1(Suppl 1):17-34. doi: 10.1038/pr.2013.204. PMID 24366461
- [Background] Hellstrom-Westas L, Rosen I. Continuous brain-function monitoring: state of the art in clinical practice. Semin Fetal Neonatal Med. 2006 Dec;11(6):503-11. doi: 10.1016/j.siny.2006.07.011. Epub 2006 Oct 24. PMID 17067863
- [Background] Hellström-Westas L, Rosén I, de Vries LS, Greisen G. Amplitude-integrated EEG Classification and Interpretation in Preterm and Term Infants. NeoReviews. 2006;7(2):e76-87.
- [Background] Shah DK, Mackay MT, Lavery S, Watson S, Harvey AS, Zempel J, Mathur A, Inder TE. Accuracy of bedside electroencephalographic monitoring in comparison with simultaneous continuous conventional electroencephalography for seizure detection in term infants. Pediatrics. 2008 Jun;121(6):1146-54. doi: 10.1542/peds.2007-1839. PMID 18519484
- [Background] Mastrangelo M, Fiocchi I, Fontana P, Gorgone G, Lista G, Belcastro V. Acute neonatal encephalopathy and seizures recurrence: a combined aEEG/EEG study. Seizure. 2013 Nov;22(9):703-7. doi: 10.1016/j.seizure.2013.05.006. Epub 2013 May 29. PMID 23725740
- [Background] Shah DK, Zempel J, Barton T, Lukas K, Inder TE. Electrographic seizures in preterm infants during the first week of life are associated with cerebral injury. Pediatr Res. 2010 Jan;67(1):102-6. doi: 10.1203/PDR.0b013e3181bf5914. PMID 19745782
- [Background] Payne ET, Zhao XY, Frndova H, McBain K, Sharma R, Hutchison JS, Hahn CD. Seizure burden is independently associated with short term outcome in critically ill children. Brain. 2014 May;137(Pt 5):1429-38. doi: 10.1093/brain/awu042. Epub 2014 Mar 4. PMID 24595203
- [Background] van Rooij LG, Toet MC, van Huffelen AC, Groenendaal F, Laan W, Zecic A, de Haan TR, van Straaten IL, Vrancken S, van Wezel G, van der Sluijs J, Ter Horst H, Gavilanes D, Laroche S, Naulaers G, de Vries LS. Effect of treatment of subclinical neonatal seizures detected with aEEG: randomized, controlled trial. Pediatrics. 2010 Feb;125(2):e358-66. doi: 10.1542/peds.2009-0136. Epub 2010 Jan 25. PMID 20100767
- [Background] Vesoulis ZA, Inder TE, Woodward LJ, Buse B, Vavasseur C, Mathur AM. Early electrographic seizures, brain injury, and neurodevelopmental risk in the very preterm infant. Pediatr Res. 2014 Apr;75(4):564-9. doi: 10.1038/pr.2013.245. Epub 2013 Dec 23. PMID 24366515
- [Background] Srinivasakumar P, Zempel J, Trivedi S, Wallendorf M, Rao R, Smith B, Inder T, Mathur AM. Treating EEG Seizures in Hypoxic Ischemic Encephalopathy: A Randomized Controlled Trial. Pediatrics. 2015 Nov;136(5):e1302-9. doi: 10.1542/peds.2014-3777. Epub 2015 Oct 19. PMID 26482675
- [Background] Hellstrom-Westas L, Rosen I, Svenningsen NW. Predictive value of early continuous amplitude integrated EEG recordings on outcome after severe birth asphyxia in full term infants. Arch Dis Child Fetal Neonatal Ed. 1995 Jan;72(1):F34-8. doi: 10.1136/fn.72.1.f34. PMID 7743282
- [Background] Thoresen M, Hellstrom-Westas L, Liu X, de Vries LS. Effect of hypothermia on amplitude-integrated electroencephalogram in infants with asphyxia. Pediatrics. 2010 Jul;126(1):e131-9. doi: 10.1542/peds.2009-2938. Epub 2010 Jun 21. PMID 20566612
- [Background] van Rooij LG, Toet MC, Osredkar D, van Huffelen AC, Groenendaal F, de Vries LS. Recovery of amplitude integrated electroencephalographic background patterns within 24 hours of perinatal asphyxia. Arch Dis Child Fetal Neonatal Ed. 2005 May;90(3):F245-51. doi: 10.1136/adc.2004.064964. PMID 15846017
- [Background] Del Rio R, Ochoa C, Alarcon A, Arnaez J, Blanco D, Garcia-Alix A. Amplitude Integrated Electroencephalogram as a Prognostic Tool in Neonates with Hypoxic-Ischemic Encephalopathy: A Systematic Review. PLoS One. 2016 Nov 1;11(11):e0165744. doi: 10.1371/journal.pone.0165744. eCollection 2016. PMID 27802300
- [Background] van Bel F, Lemmers P, Naulaers G. Monitoring neonatal regional cerebral oxygen saturation in clinical practice: value and pitfalls. Neonatology. 2008;94(4):237-44. doi: 10.1159/000151642. Epub 2008 Sep 11. PMID 18784420
- [Background] Alderliesten T, De Vis JB, Lemmers PM, Hendrikse J, Groenendaal F, van Bel F, Benders MJ, Petersen ET. Brain oxygen saturation assessment in neonates using T2-prepared blood imaging of oxygen saturation and near-infrared spectroscopy. J Cereb Blood Flow Metab. 2017 Mar;37(3):902-913. doi: 10.1177/0271678X16647737. Epub 2016 Jul 20. PMID 27151900
- [Background] Chock VY, Rose LA, Mante JV, Punn R. Near-infrared spectroscopy for detection of a significant patent ductus arteriosus. Pediatr Res. 2016 Nov;80(5):675-680. doi: 10.1038/pr.2016.148. Epub 2016 Sep 7. PMID 27603562
- [Background] Hall RW, Hall-Barrow J, Garcia-Rill E. Neonatal regionalization through telemedicine using a community-based research and education core facility. Ethn Dis. 2010 Winter;20(1 Suppl 1):S1-136-40. PMID 20521402
- [Background] Burke BL Jr, Hall RW; SECTION ON TELEHEALTH CARE. Telemedicine: Pediatric Applications. Pediatrics. 2015 Jul;136(1):e293-308. doi: 10.1542/peds.2015-1517. PMID 26122813
- [Background] McConnochie K, Wood N, Herendeen N, ten Hoopen C, Denk L, Neuderfer J. Integrating telemedicine in urban pediatric primary care: provider perspectives and performance. Telemed J E Health. 2010 Apr;16(3):280-8. doi: 10.1089/tmj.2009.0112. PMID 20406114
- [Background] Variane GF, Cunha LM, Pinto P, Brandao P, Mascaretti RS, Magalhaes M, Sant'Anna GM. Therapeutic Hypothermia in Brazil: A MultiProfessional National Survey. Am J Perinatol. 2019 Sep;36(11):1150-1156. doi: 10.1055/s-0038-1676052. Epub 2018 Dec 15. PMID 30553235
- [Background] Triulzi F, Parazzini C, Righini A. Patterns of damage in the mature neonatal brain. Pediatr Radiol. 2006 Jul;36(7):608-20. doi: 10.1007/s00247-006-0203-5. Epub 2006 May 18. PMID 16770665
- [Background] Ferriero DM. Neonatal brain injury. N Engl J Med. 2004 Nov 4;351(19):1985-95. doi: 10.1056/NEJMra041996. No abstract available. PMID 15525724
- [Background] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433
- [Background] Abend NS, Wusthoff CJ, Goldberg EM, Dlugos DJ. Electrographic seizures and status epilepticus in critically ill children and neonates with encephalopathy. Lancet Neurol. 2013 Dec;12(12):1170-9. doi: 10.1016/S1474-4422(13)70246-1. PMID 24229615
- [Background] Murray DM, Boylan GB, Ali I, Ryan CA, Murphy BP, Connolly S. Defining the gap between electrographic seizure burden, clinical expression and staff recognition of neonatal seizures. Arch Dis Child Fetal Neonatal Ed. 2008 May;93(3):F187-91. doi: 10.1136/adc.2005.086314. Epub 2007 Jul 11. PMID 17626147
- [Background] Burnett AC, Cheong JLY, Doyle LW. Biological and Social Influences on the Neurodevelopmental Outcomes of Preterm Infants. Clin Perinatol. 2018 Sep;45(3):485-500. doi: 10.1016/j.clp.2018.05.005. PMID 30144851
- [Background] Joseph RM, O'Shea TM, Allred EN, Heeren T, Hirtz D, Jara H, Leviton A, Kuban KC; ELGAN Study Investigators. Neurocognitive and Academic Outcomes at Age 10 Years of Extremely Preterm Newborns. Pediatrics. 2016 Apr;137(4):e20154343. doi: 10.1542/peds.2015-4343. Epub 2016 Mar 22. PMID 27006473
- [Background] Cheong JL, Doyle LW, Burnett AC, Lee KJ, Walsh JM, Potter CR, Treyvaud K, Thompson DK, Olsen JE, Anderson PJ, Spittle AJ. Association Between Moderate and Late Preterm Birth and Neurodevelopment and Social-Emotional Development at Age 2 Years. JAMA Pediatr. 2017 Apr 3;171(4):e164805. doi: 10.1001/jamapediatrics.2016.4805. Epub 2017 Apr 3. PMID 28152144
- [Background] Bosi G, Garani G, Scorrano M, Calzolari E; IMER Working Party. Temporal variability in birth prevalence of congenital heart defects as recorded by a general birth defects registry. J Pediatr. 2003 Jun;142(6):690-8. doi: 10.1067/mpd.2003.243. PMID 12838199
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541
- [Background] Dimitropoulos A, McQuillen PS, Sethi V, Moosa A, Chau V, Xu D, Brant R, Azakie A, Campbell A, Barkovich AJ, Poskitt KJ, Miller SP. Brain injury and development in newborns with critical congenital heart disease. Neurology. 2013 Jul 16;81(3):241-8. doi: 10.1212/WNL.0b013e31829bfdcf. Epub 2013 Jun 14. PMID 23771484
- [Background] Limperopoulos C, Majnemer A, Shevell MI, Rosenblatt B, Rohlicek C, Tchervenkov C. Neurologic status of newborns with congenital heart defects before open heart surgery. Pediatrics. 1999 Feb;103(2):402-8. doi: 10.1542/peds.103.2.402. PMID 9925832
- [Background] Gunn JK, Beca J, Hunt RW, Olischar M, Shekerdemian LS. Perioperative amplitude-integrated EEG and neurodevelopment in infants with congenital heart disease. Intensive Care Med. 2012 Sep;38(9):1539-47. doi: 10.1007/s00134-012-2608-y. Epub 2012 Jun 1. PMID 22653373
- [Background] Gunn JK, Beca J, Penny DJ, Horton SB, d'Udekem YA, Brizard CP, Finucane K, Olischar M, Hunt RW, Shekerdemian LS. Amplitude-integrated electroencephalography and brain injury in infants undergoing Norwood-type operations. Ann Thorac Surg. 2012 Jan;93(1):170-6. doi: 10.1016/j.athoracsur.2011.08.014. Epub 2011 Nov 9. PMID 22075220
- [Background] Toso PA, Gonzalez AJ, Perez ME, Kattan J, Fabres JG, Tapia JL, Gonzalez HS. Clinical utility of early amplitude integrated EEG in monitoring term newborns at risk of neurological injury. J Pediatr (Rio J). 2014 Mar-Apr;90(2):143-8. doi: 10.1016/j.jped.2013.07.004. Epub 2013 Oct 30. PMID 24184304
- [Background] Shah NA, Wusthoff CJ. How to use: amplitude-integrated EEG (aEEG). Arch Dis Child Educ Pract Ed. 2015 Apr;100(2):75-81. doi: 10.1136/archdischild-2013-305676. Epub 2014 Jul 17. PMID 25035312
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Background] Simbruner G, Mittal RA, Rohlmann F, Muche R; neo.nEURO.network Trial Participants. Systemic hypothermia after neonatal encephalopathy: outcomes of neo.nEURO.network RCT. Pediatrics. 2010 Oct;126(4):e771-8. doi: 10.1542/peds.2009-2441. Epub 2010 Sep 20. PMID 20855387
- [Background] Skranes JH, Lohaugen G, Schumacher EM, Osredkar D, Server A, Cowan FM, Stiris T, Fugelseth D, Thoresen M. Amplitude-Integrated Electroencephalography Improves the Identification of Infants with Encephalopathy for Therapeutic Hypothermia and Predicts Neurodevelopmental Outcomes at 2 Years of Age. J Pediatr. 2017 Aug;187:34-42. doi: 10.1016/j.jpeds.2017.04.041. Epub 2017 May 23. PMID 28549636
- [Background] Sarkar S, Barks JD, Donn SM. Should amplitude-integrated electroencephalography be used to identify infants suitable for hypothermic neuroprotection? J Perinatol. 2008 Feb;28(2):117-22. doi: 10.1038/sj.jp.7211882. Epub 2007 Nov 15. PMID 18004390
- [Background] Chandrasekaran M, Chaban B, Montaldo P, Thayyil S. Predictive value of amplitude-integrated EEG (aEEG) after rescue hypothermic neuroprotection for hypoxic ischemic encephalopathy: a meta-analysis. J Perinatol. 2017 Jun;37(6):684-689. doi: 10.1038/jp.2017.14. Epub 2017 Mar 2. PMID 28252661
- [Background] Ancora G, Maranella E, Grandi S, Sbravati F, Coccolini E, Savini S, Faldella G. Early predictors of short term neurodevelopmental outcome in asphyxiated cooled infants. A combined brain amplitude integrated electroencephalography and near infrared spectroscopy study. Brain Dev. 2013 Jan;35(1):26-31. doi: 10.1016/j.braindev.2011.09.008. Epub 2011 Nov 13. PMID 22082686
- [Background] Jain SV, Pagano L, Gillam-Krakauer M, Slaughter JC, Pruthi S, Engelhardt B. Cerebral regional oxygen saturation trends in infants with hypoxic-ischemic encephalopathy. Early Hum Dev. 2017 Oct;113:55-61. doi: 10.1016/j.earlhumdev.2017.07.008. Epub 2017 Aug 1. PMID 28772198
- [Background] Lemmers PM, Zwanenburg RJ, Benders MJ, de Vries LS, Groenendaal F, van Bel F, Toet MC. Cerebral oxygenation and brain activity after perinatal asphyxia: does hypothermia change their prognostic value? Pediatr Res. 2013 Aug;74(2):180-5. doi: 10.1038/pr.2013.84. Epub 2013 May 31. PMID 23728382
- [Background] Tekgul H, Gauvreau K, Soul J, Murphy L, Robertson R, Stewart J, Volpe J, Bourgeois B, du Plessis AJ. The current etiologic profile and neurodevelopmental outcome of seizures in term newborn infants. Pediatrics. 2006 Apr;117(4):1270-80. doi: 10.1542/peds.2005-1178. PMID 16585324
- [Background] Hellstrom-Westas L, Rosen I, Svenningsen NW. Cerebral function monitoring during the first week of life in extremely small low birthweight (ESLBW) infants. Neuropediatrics. 1991 Feb;22(1):27-32. doi: 10.1055/s-2008-1071411. PMID 2038424
- [Background] Wikstrom S, Pupp IH, Rosen I, Norman E, Fellman V, Ley D, Hellstrom-Westas L. Early single-channel aEEG/EEG predicts outcome in very preterm infants. Acta Paediatr. 2012 Jul;101(7):719-26. doi: 10.1111/j.1651-2227.2012.02677.x. Epub 2012 Apr 24. PMID 22530996
- [Background] Soubasi V, Mitsakis K, Sarafidis K, Griva M, Nakas CT, Drossou V. Early abnormal amplitude-integrated electroencephalography (aEEG) is associated with adverse short-term outcome in premature infants. Eur J Paediatr Neurol. 2012 Nov;16(6):625-30. doi: 10.1016/j.ejpn.2012.02.008. Epub 2012 Mar 15. PMID 22425390
- [Background] Klebermass K, Olischar M, Waldhoer T, Fuiko R, Pollak A, Weninger M. Amplitude-integrated EEG pattern predicts further outcome in preterm infants. Pediatr Res. 2011 Jul;70(1):102-8. doi: 10.1203/PDR.0b013e31821ba200. PMID 21436758
- [Background] Variane GFT, Magalhaes M, Gasperine R, Alves HCBR, Scoppetta TLPD, Figueredo RJG, Rodrigues FPM, Netto A, Mimica MJ, Gallacci CB. Early amplitude-integrated electroencephalography for monitoring neonates at high risk for brain injury. J Pediatr (Rio J). 2017 Sep-Oct;93(5):460-466. doi: 10.1016/j.jped.2016.12.003. Epub 2017 Feb 23. PMID 28238681
- [Background] Hyttel-Sorensen S, Pellicer A, Alderliesten T, Austin T, van Bel F, Benders M, Claris O, Dempsey E, Franz AR, Fumagalli M, Gluud C, Grevstad B, Hagmann C, Lemmers P, van Oeveren W, Pichler G, Plomgaard AM, Riera J, Sanchez L, Winkel P, Wolf M, Greisen G. Cerebral near infrared spectroscopy oximetry in extremely preterm infants: phase II randomised clinical trial. BMJ. 2015 Jan 5;350:g7635. doi: 10.1136/bmj.g7635. PMID 25569128
- [Background] Lemmers PM, Toet MC, van Bel F. Impact of patent ductus arteriosus and subsequent therapy with indomethacin on cerebral oxygenation in preterm infants. Pediatrics. 2008 Jan;121(1):142-7. doi: 10.1542/peds.2007-0925. PMID 18166568
- [Background] Underwood MA, Milstein JM, Sherman MP. Near-infrared spectroscopy as a screening tool for patent ductus arteriosus in extremely low birth weight infants. Neonatology. 2007;91(2):134-9. doi: 10.1159/000097131. Epub 2006 Nov 20. PMID 17344664
- [Background] Olischar M, Shany E, Aygun C, Azzopardi D, Hunt RW, Toet MC, Hamosh A, de Vries LS, Hellstrom-Westas L, Theda C. Amplitude-integrated electroencephalography in newborns with inborn errors of metabolism. Neonatology. 2012;102(3):203-11. doi: 10.1159/000339567. Epub 2012 Jul 12. PMID 22797054
- [Background] Helderman JB, Welch CD, Leng X, O'Shea TM. Sepsis-associated electroencephalographic changes in extremely low gestational age neonates. Early Hum Dev. 2010 Aug;86(8):509-13. doi: 10.1016/j.earlhumdev.2010.06.006. Epub 2010 Aug 12. PMID 20708356
- [Background] ter Horst HJ, Mud M, Roofthooft MT, Bos AF. Amplitude integrated electroencephalographic activity in infants with congenital heart disease before surgery. Early Hum Dev. 2010 Dec;86(12):759-64. doi: 10.1016/j.earlhumdev.2010.08.028. PMID 20970264
- [Background] Latal B, Wohlrab G, Brotschi B, Beck I, Knirsch W, Bernet V. Postoperative Amplitude-Integrated Electroencephalography Predicts Four-Year Neurodevelopmental Outcome in Children with Complex Congenital Heart Disease. J Pediatr. 2016 Nov;178:55-60.e1. doi: 10.1016/j.jpeds.2016.06.050. Epub 2016 Jul 22. PMID 27453368
- [Background] Dodge-Khatami J, Gottschalk U, Eulenburg C, Wendt U, Schnegg C, Rebel M, Reichenspurner H, Dodge-Khatami A. Prognostic value of perioperative near-infrared spectroscopy during neonatal and infant congenital heart surgery for adverse in-hospital clinical events. World J Pediatr Congenit Heart Surg. 2012 Apr 1;3(2):221-8. doi: 10.1177/2150135111426298. PMID 23804778
- [Background] Colasacco C, Worthen M, Peterson B, Lamberti J, Spear R. Near-infrared spectroscopy monitoring to predict postoperative renal insufficiency following repair of congenital heart disease. World J Pediatr Congenit Heart Surg. 2011 Oct 1;2(4):536-40. doi: 10.1177/2150135111411932. PMID 23804464
- [Background] Hoffman GM, Ghanayem NS, Scott JP, Tweddell JS, Mitchell ME, Mussatto KA. Postoperative Cerebral and Somatic Near-Infrared Spectroscopy Saturations and Outcome in Hypoplastic Left Heart Syndrome. Ann Thorac Surg. 2017 May;103(5):1527-1535. doi: 10.1016/j.athoracsur.2016.09.100. Epub 2016 Dec 21. PMID 28012642
- [Background] Clair MP, Rambaud J, Flahault A, Guedj R, Guilbert J, Guellec I, Durandy A, Demoulin M, Jean S, Mitanchez D, Chalard F, Sileo C, Carbajal R, Renolleau S, Leger PL. Prognostic value of cerebral tissue oxygen saturation during neonatal extracorporeal membrane oxygenation. PLoS One. 2017 Mar 9;12(3):e0172991. doi: 10.1371/journal.pone.0172991. eCollection 2017. PMID 28278259
- [Background] Sood BG, McLaughlin K, Cortez J. Near-infrared spectroscopy: applications in neonates. Semin Fetal Neonatal Med. 2015 Jun;20(3):164-72. doi: 10.1016/j.siny.2015.03.008. Epub 2015 Apr 29. PMID 25934116
- [Background] Johnson BA, Hoffman GM, Tweddell JS, Cava JR, Basir M, Mitchell ME, Scanlon MC, Mussatto KA, Ghanayem NS. Near-infrared spectroscopy in neonates before palliation of hypoplastic left heart syndrome. Ann Thorac Surg. 2009 Feb;87(2):571-7; discussion 577-9. doi: 10.1016/j.athoracsur.2008.10.043. PMID 19161781
- [Background] Hanson SJ, Berens RJ, Havens PL, Kim MK, Hoffman GM. Effect of volume resuscitation on regional perfusion in dehydrated pediatric patients as measured by two-site near-infrared spectroscopy. Pediatr Emerg Care. 2009 Mar;25(3):150-3. doi: 10.1097/PEC.0b013e31819a7f60. PMID 19262423
- [Background] Pichler G, Holler N, Baik-Schneditz N, Schwaberger B, Mileder L, Stadler J, Avian A, Pansy J, Urlesberger B. Avoiding Arterial Hypotension in Preterm Neonates (AHIP)-A Single Center Randomised Controlled Study Investigating Simultaneous Near Infrared Spectroscopy Measurements of Cerebral and Peripheral Regional Tissue Oxygenation and Dedicated Interventions. Front Pediatr. 2018 Feb 1;6:15. doi: 10.3389/fped.2018.00015. eCollection 2018. PMID 29450194
- [Background] Variane GFT, Chock VY, Netto A, Pietrobom RFR, Van Meurs KP. Simultaneous Near-Infrared Spectroscopy (NIRS) and Amplitude-Integrated Electroencephalography (aEEG): Dual Use of Brain Monitoring Techniques Improves Our Understanding of Physiology. Front Pediatr. 2020 Jan 21;7:560. doi: 10.3389/fped.2019.00560. eCollection 2019. PMID 32039117
- [Background] Pauliah SS, Shankaran S, Wade A, Cady EB, Thayyil S. Therapeutic hypothermia for neonatal encephalopathy in low- and middle-income countries: a systematic review and meta-analysis. PLoS One. 2013;8(3):e58834. doi: 10.1371/journal.pone.0058834. Epub 2013 Mar 19. PMID 23527034
- [Background] Frenkel N, Friger M, Meledin I, Berger I, Marks K, Bassan H, Shany E. Neonatal seizure recognition--comparative study of continuous-amplitude integrated EEG versus short conventional EEG recordings. Clin Neurophysiol. 2011 Jun;122(6):1091-7. doi: 10.1016/j.clinph.2010.09.028. Epub 2011 Jan 7. PMID 21216190
- [Background] Rakshasbhuvankar A, Paul S, Nagarajan L, Ghosh S, Rao S. Amplitude-integrated EEG for detection of neonatal seizures: a systematic review. Seizure. 2015 Dec;33:90-8. doi: 10.1016/j.seizure.2015.09.014. Epub 2015 Sep 26. PMID 26456517
- [Background] Udeh C, Udeh B, Rahman N, Canfield C, Campbell J, Hata JS. Telemedicine/Virtual ICU: Where Are We and Where Are We Going? Methodist Debakey Cardiovasc J. 2018 Apr-Jun;14(2):126-133. doi: 10.14797/mdcj-14-2-126. PMID 29977469
- [Background] Kahn JM, Le TQ, Barnato AE, Hravnak M, Kuza CC, Pike F, Angus DC. ICU Telemedicine and Critical Care Mortality: A National Effectiveness Study. Med Care. 2016 Mar;54(3):319-25. doi: 10.1097/MLR.0000000000000485. PMID 26765148
- [Background] Maldonado JM, Marques AB, Cruz A. Telemedicine: challenges to dissemination in Brazil. Cad Saude Publica. 2016 Nov 3;32Suppl 2(Suppl 2):e00155615. doi: 10.1590/0102-311X00155615. English, Portuguese. PMID 27828681
- [Derived] Variane GFT, Magalhaes M, Pietrobom RFR, Netto A, Rodrigues DP, Gasperini R, Sant'Anna GM. Protecting brains and saving futures guidelines: A prospective, multicenter, and observational study on the use of telemedicine for neonatal neurocritical care in Brazil. PLoS One. 2022 Jan 12;17(1):e0262581. doi: 10.1371/journal.pone.0262581. eCollection 2022. PMID 35020756
- See also: 25. World Health Organization. A health telematics policy in support of WHO's Health-for-All Strategy for Global Health Development. Geneva (Switzerland); 1998. — https://apps.who.int/iris/handle/10665/63857
- See also: 26. World Health Organization. Telemedicine: Opportunities and Development in Member States: Report on the second global survey on eHealth. Geneva (Switzerland); 2010. — https://apps.who.int/iris/handle/10665/44497
- See also: 30. Ministério da Saúde. DATASUS. [online] Tabnet. [accessed on Jan 10th 2018] — https://datasus.saude.gov.br/informacoes-de-saude-tabnet/